CLINICAL TRIAL: NCT06426225
Title: Should General Anesthesia or Spinal Aneshtesia With Ketofol Sedation Be Applied in Umblical Hernia Operations ?
Brief Title: Spinal Or General Anesthesia For Umblical Hernia Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Nargiz Mammadova, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1646
Record Dates: First submitted 2024-05-07; First posted 2024-05-23 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Umbilical Hernia; Spinal Aneshtesia; General Anesthesia
MeSH Terms: conditions — Hernia, Umbilical | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Anesthesia (Active Comparator): As premedication 0.03mg/kg midazolam was administered. During general anesthesia, 3 mg/kg propofol, 0.6 mg/kg rocuronium and 1 mcg/kg fentanyl were administered to all patients for induction.
  Interventions: Other: General Anesthesia
- Spinal Anesthesia (Active Comparator): As premedication 0.03mg/kg midazolam was administered. After premedication Spinal Anesthesia applied. Group will be sedated with ketofol after spinal anesthesia. Ketamine:propofol mixture will be prepared as 1:1 5mg/ml propofol and 5mg/ml ketamine. Surgery will begin when the Ramsey sedation scale reaches 3.
  Interventions: Other: Spinal Aneshtesia

INTERVENTIONS:
Other: General Anesthesia — General Anesthesia Applied Group 2 Patients.
  Arms: General Anesthesia
Other: Spinal Aneshtesia — Spinal Anesthesia and Ketofol Sedation Applied Group 1 Patients.
  Arms: Spinal Anesthesia

SUMMARY:
In this study, the investigators compared spinal anesthesia under ketofol (ketamine-propofol combination) sedation with general anesthesia in terms of intraoperative and postoperative hemodynamics, respiratory parameters and cost in patients undergoing umbilical hernia operation. the investigator aimed to provide the most appropriate and hemodynamically stable option for the patient, to decrease the complication rates and to reduce the associated costs.

DETAILED DESCRIPTION:
This study was carried out at the Ministry of Health Ankara City Hospital Operating Room, after receiving ethics committee approval.Preoperative evaluation was performed before the operation in cases undergoing elective umbilical hernia surgery.Complications and side effects are explained in detail.Verbal and written consents were obtained from the subjects who agreed to participate in the study.In patients undergoing umbilical hernia surgery, general anesthesia and spinal anesthesia under propofol and ketamine (ketamine-propofol combination) sedation were compared in terms of intraoperative and postoperative hemodynamics, aldrete score, pain score, respiratory parameters, and cost. The patients, who had fasted for 8 hours before the operation, were taken to the operating room without premedication.

In all cases, a peripheral venous catheter cannulated on the dorsal part of the hand (20G, Plusflon i.v. Cannula, India) .Standard monitoring was applied.

Group1. As premedication 0.03mg/kg midazolam was administered . For spinal anesthesia, 15 mg heavy-bupivacaine, sedation was provided with ketofol.

ketamine:propofol mixture was prepared as 1:1 5mg/ml propofol and 5mg/ml ketamine

1 mg/kg ketofol administered i.v. Group2 . As premedication 0.03mg/kg midazolam was administered.In general anesthesia to all patients after induction 3 mg/kg propofol, 0.6 mg/kg rocuronium and 1 mcg/kg fentanyl Bispectral index and non-invasive blood pressure was monitored, a urinary catheter was placed. Anesthesia was maintained with sevoflurane and fentanyl to keep BIS values between 40-60.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients between the ages of 18 and 65 who would undergo Umbilical hernia surgery were included in the study.

Exclusion Criteria:

* who do not accept the procedure
* serious cardiovasculer disease ,renal, hematological (bleeding diathesis, under anticoagulant therapy, those with hemoglobin value below 10 g/dl) disease, hepatic disease, cerebrovascular, neurological or psychiatric diseases,
* those who are contraindicated for spinal anesthesia,
* Those who are allergic to one of the local anesthetics to be used, with drug and alcohol addiction,
* pregnant or breastfeeding
* using drugs and analgesics effective on the central nervous system were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Heart Rate | preoperative 0. minute, intraoperative 10.minute, intraoperative 20.minute, intraoperative 30.minute, Postoperative 0.minute, Postoperative 10.minute, Postoperative 20.minute, Postoperative 30.minute
  During Perioperative Period Heart rate was measured
systolic blood pressure | preoperative 0. minute, intraoperative 10.minute, intraoperative 20.minute, intraoperative 30.minute, Postoperative 0.minute, Postoperative 10.minute, Postoperative 20.minute, Postoperative 30.minute
  non invasive blood pressure measurement
diastolic blood pressure | preoperative 0. minute, intraoperative 10.minute, intraoperative 20.minute, intraoperative 30.minute, Postoperative 0.minute, Postoperative 10.minute, Postoperative 20.minute, Postoperative 30.minute
  non invasive blood pressure measurement
mean arterial blood pressure | preoperative 0. minute, intraoperative 10.minute, intraoperative 20.minute, intraoperative 30.minute, Postoperative 0.minute, Postoperative 10.minute, Postoperative 20.minute, Postoperative 30.minute
  non invasive blood pressure measurement
hospital stay | From hospital admission to discharge
  Length of hospital stay was recorded.
Cost | From hospital admission to discharge
  Bill amount during hospitalization

SECONDARY OUTCOMES:
Postoperative NRS | Postoperative 30.minute, Postoperative 12. hour
  postoperative numeric rating scale was evaluated, 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable
Postoperative Aldrete Score | Postoperative first 1 hour
  Postoperative Aldrete score was evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] KROBOT, R. i PREMUŽIĆ, J. (2013). Comparison of general and spinal anaesthesia in patients undergoing open ventral hernia repair. Periodicum biologorum, 115 (2), 225-229. Preuzeto s https://hrcak.srce.hr/105984
- [Background] Germano P, Siboni S, Milito P, Mautone G, Resta M, Bonavina L. Ventral hernia repair under neuraxial anesthesia. Eur Surg. 2022;54(1):54-58. doi: 10.1007/s10353-021-00731-x. Epub 2021 Jul 20. PMID 34306042